CLINICAL TRIAL: NCT04467528
Title: Efficacy of Electroacupuncture as an Adjunctive Treatment in Gastrointestinal Motility in Patients After Abdominal Surgery
Brief Title: Electroacupuncture for Gastrointestinal Dysmotility After Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH109-REC3-040
Record Dates: First submitted 2020-05-20; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Abdominal Surgery
Keywords: abdominal surgery; acupuncture; electroacupuncture
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture combined with conventional drug therapy (Experimental): Conventional drug therapy:
  All participants receive intravenous infusion of metoclopramide(10mg) every 12 hours in the trial
  For participants with abdominal distension:
  Electroacupuncture will be applied to the acupoints (LI4, PC6, ST36, SP6) 30min
  For participants with post-operative ileus:
  Electroacupuncture will be applied to the acupoints (LI4, SJ6, ST36, ST37) 30min
  32# acupuncture needle used and twice daily for three days
  Interventions: Device: Electroacupuncture; Drug: Conventional drug therapy
- Conventional drug therapy (Active Comparator): Conventional drug therapy:
  All participants receive intravenous infusion of metoclopramide(10mg) every 12 hours in the trial
  Interventions: Drug: Conventional drug therapy

INTERVENTIONS:
Device: Electroacupuncture — Experimental: Electroacupuncture combined with conventional drug therapy
  Conventional drug therapy:
  All participants receive intravenous infusion of metoclopramide(10mg) every 12 hours in the trial
  For participants with abdominal distension:
  Electroacupuncture will be applied to the acupoints (LI4, PC6, ST36, SP6) 30min
  For participants with post-operative ileus:
  Electroacupuncture will be applied to the acupoints (LI4, SJ6, ST36, ST37) 30min
  32# acupuncture needle used and twice daily for three days
  Arms: Electroacupuncture combined with conventional drug therapy
Drug: Conventional drug therapy — Conventional drug therapy:
  All participants receive intravenous infusion of metoclopramide(10mg) every 12 hours in the trial

SUMMARY:
In Taiwan, the number of patients who underwent abdominal surgery that attributed to gastrointestinal diseases, gynecological diseases, and cancer is increasing. Practically, some of the patients have unsatisfactory response to conventional medical treatment, which result in abnormal gastrointestinal function, prolonged bedtime, and increased hospital stay, as well as an increased risk of infection. Therefore, search for an effective and safe treatment that could be integrated to current medical treatment is of importance in the care of such patients.

Being with a long period of clinical experience and evidence-based curative effect, acupuncture could be applied as an adjunctive treatment for the complications of abdominal surgery. Currently, this patient-centered, pragmatic clinical trial compares the efficacy of using conventional medication alone and a combination of electroacupuncture and conventional drugs. The aim of this study is trying to explore acceptable and beneficial strategy to reduce the clinical symptoms, to improve quality of life, and decrease medical expenses.

DETAILED DESCRIPTION:
A total of 80 volunteers of patients underwent abdominal surgery will be recruited from the intensive care unit of China Medical University Hospital. After diagnosis by surgeon, these patients will be assigned to receive the conventional drug alone or the conventional drug combined electroacupuncture treatment. All participants receive intravenous injection the conventional drug, Metoclopramide, every 12 hours in the trial. Electroacupuncture, twice daily for three days, is administered 48-72 hours after abdominal surgery. Visual analogue scale, feeding volume, gastric residual volume and assessment of adverse events will be done for every visit. Laboratory biochemistry analysis and other assessments including Visual Analogue Scale, Acute Physiology and Chronic Health Evaluation II score, and Sequential Organ Failure Assessment score will be completed at baseline and the end of intervention(3 days after initation of the intervention). Physiological and operative severity scores for the enumeration of mortality and morbidity (POSSUM) score will be done at the baseline. Instrumental examinations including heart rate variability and traditional Chinese medicine four examinations will be given before and after intervention. We expect that the efficacy of combined electroacupuncture with conventional drug is superior to conventional drug only in alleviation of gastrointestinal distension or/and improvement of motility in patients who underwent abdominal surgery. Moreover, we will further speculate the mechanism by analyzing laboratory data.

ELIGIBILITY:
Inclusion Criteria:

1. more than 20 years old.
2. Underwent abdominal surgery within one month
3. Meet one or both of the following indications

   1. Participants have abdominal distension after abdominal surgery which affects gastrointestinal motility. After medical treatment, the visual pain scale score remained above three points
   2. Participants have post-operative ileus after abdominal surgery. After medical treatment, the gastric residual volume is still greater than 300 ml under the intestinal nutrition support
4. Had signed the informed consent with fully understand the aim of the clinical trial

Exclusion Criteria:

1. Hemorrhagic disease or coagulation dysfunction
2. Local skin infection
3. Fear of needles or electrical stimulation
4. Any severe chronic or uncontrollable complications

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | baseline, 1st day of the intervention, 2nd day of the intervention, 3rd day of the intervention
  Changes from baseline to 1st day of the intervention, 2nd day of the intervention, 3rd day of the intervention
Daily feeding volume | baseline, 1st day of the intervention, 2nd day of the intervention, 3rd day of the intervention
  Changes from baseline to 1st day of the intervention, 2nd day of the intervention, 3rd day of the intervention
Gastric residual volume | baseline, 1st day of the intervention, 2nd day of the intervention, 3rd day of the intervention
  Changes from baseline to 1st day of the intervention, 2nd day of the intervention, 3rd day of the intervention

SECONDARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation II score | baseline, Day 3 of the intervention
  Changes from baseline to 3rd day of the intervention
Sequential Organ Failure Assessment score | baseline, Day 3 of the intervention
  Changes from baseline to 3rd day of the intervention
Physiological and operative severity scores for the enumeration of mortality and morbidity score | baseline
  To predict morbidity and mortality of the patients in ICU
Blood examination | baseline, Day 3 of the intervention
  Changes of CBC, ALT, AST, BUN, Creatinine, CRP from baseline to 3rd day of the intervention
Laboratory examination | baseline, Day 3 of the intervention
  Changes of cytokines (IL-1,6,10,12) from baseline to 3rd day of the intervention
Heart rate variability | baseline, 1st day of the intervention, 2nd day of the intervention, 3rd day of the intervention
  Changes from baseline to 1st day of the intervention, 2nd day of the intervention, 3rd day of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Cheng Huang, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No